CLINICAL TRIAL: NCT02684162
Title: A Phase II Trial to Assess the Efficacy and Toxicity of SGI-110 With DLI for the Treatment of AML or MDS Relapsing After Allogeneic Stem Cell Transplantation
Brief Title: Guadecitabine and Donor Lymphocyte Infusion in Treating Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome Relapsing After Allogeneic Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0117; NCI-2016-00343 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0117 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-02-12; First posted 2016-02-17 (Estimated); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Recurrent Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (guadecitabine, DLI) (Experimental): Patients receive guadecitabine SC QD on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive DLI IV over 10-30 minutes on day 6 of cycles 2, 4, and 6 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Donor Lymphocytes; Drug: Guadecitabine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Donor Lymphocytes — Given IV
Drug: Guadecitabine — Given SC
  Other Names: DNMT inhibitor SGI-110; S110; SGI-110
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase IIa trial studies how well guadecitabine works in treating patients with acute myelogenous leukemia and myelodysplastic syndrome that has returned after a period of improvement after allogeneic stem cell transplant. Guadecitabine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft-versus-host disease). Giving guadecitabine before the transplant may stop this from happening. Once the donated stem cells begin working, the patient's immune system may see the remaining cancer cells as not belonging in the patient's body and destroy them. Giving an infusion of the donor's white blood cells (donor lymphocyte infusion) may boost this effect.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete response (CR) rate of guadecitabine (SGI-110) with or without donor lymphocyte infusion (DLI) either for the treatment of morphologic relapse or the presence of minimal residual disease (MRD) in patients with acute myeloid leukemia or myelodysplastic syndrome after hematopoietic stem cell transplantation in patients with AML and MDS (cohort 1 and 2).

II. The relapse-free survival with the use of SGI-110 as maintenance therapy in patients with high risk acute myeloid leukemia or myelodysplastic syndrome after hematopoietic stem cell transplantation (cohort 3).

SECONDARY OBJECTIVES:

I. To determine the safety and toxicity of SGI-110 with or without DLI in this subject population.

II. To evaluate overall response and survival.

OUTLINE:

Patients receive guadecitabine subcutaneously (SC) once daily (QD) on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive DLI intravenously (IV) over 10-30 minutes on day 6 of cycles 2, 4, and 6 in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) and myelodysplastic syndrome (including chronic myelomonocytic leukemia [CMML]) according to WHO classification that underwent first allogeneic hematopoietic cell transplant (HSCT) with either peripheral blood or bone marrow as the source of the hematopoietic stem cells
* No more than 1 antigen mismatch at human leukocyte antigen (HLA)-A, B, C, DRB1 and DQB1 locus for either related or unrelated donor
* High risk AML and MDS patients will be included
* Cohort 1: morphological relapse after stem cell transplant:

  * MDS patients: re-appearance of dysplastic changes in the bone marrow, with or without increase in bone marrow last count, which is pathologically consistent with myelodysplastic syndrome;
  * AML patients: bone marrow blast count >= 5%
* Cohort 2: Persistence or reappearance of minimal residual disease by flow cytometry or cytogenetic or molecular testing while being in morphological remission after allogeneic stem cell transplantation
* Cohort 3: High risk AML and MDS patients who are in complete remission morphologically with no evidence of minimal residual disease by flow cytometry or cytogenetic or molecular testing after allogeneic stem cell transplantation
* MDS patients:

  * Cytogenetics consistent with poor or very poor risk group by 5-risk classification;
  * Cytogenetics consistent with monosomal karyotype
  * Bone marrow blast count > 5% but less than 20% at any time during their disease course before HSCT
  * Peripheral blood blast =< 5% at HSCT
  * Therapy-related MDS
* AML patients:

  * Cytogenetics and molecular features consistent with adverse risk group by European LeukemiaNet classification for AML;
  * Presence of minimal residual disease by multi-color flow cytometry or cytogenetics or molecular studies at the time of HSCT;
  * Presence of active disease defined as bone marrow blast count > 5% but less than =< 10% at the time of HSCT
  * Peripheral blood blast count =< 5% at HSCT
  * Therapy-related AML
* Be able to start the drug therapy between 42 to 100 days following allogeneic SCT;

  * No more than 1 prior allogeneic SCT
  * Post-transplant bone marrow consistent with complete remission with no evidence of minimal residual disease by flow-cytometry or cytogenetics or molecular testing
  * Adequate engraftment within 14 days prior to starting study drug: absolute neutrophil count (ANC) >= 1.0 x 10^9/L without daily use of myeloid growth factor; and, platelet >= 50 x 10^9/L without platelet transfusion within 1 week
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Serum creatinine =< 1.5 mg/dL or creatinine clearance greater or equal than 40 cc/min as defined by the Cockcroft-Gault equation
* Serum bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate transaminase (aspartate aminotransferase [AST]) or alanine transaminase (alanine aminotransferase [ALT]) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x upper limit (UL)
* No active bleeding
* No uncontrolled graft versus host disease (GVHD)
* No clinical evidence of life-threatening infection
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
* Human immunodeficiency virus (HIV) negative and hepatitis B surface antigen (HBs-Ag) negative
* Negative serum or urine pregnancy test for women with reproductive potential; the only subjects who will be exempt from this criterion are postmenopausal women (defined as women who have been amenorrheic for > 12 months) or subjects who have been surgically sterilized or otherwise proven sterile

Exclusion Criteria:

* Use of any anti-leukemic agents after relapse is documented (note that the use of these anti-leukemic agents given as post-transplant maintenance therapy is allowed in this study, e.g., subcutaneous or oral 5-azacytidine or FLT3 inhibitors for maintenance) for cohorts 1 and 2
* Bone marrow blast count > 60% for cohort 1
* Use of any of the following after transplantation and prior to starting study therapy for cohort 3:

  * Investigational agents/therapies
  * Anti-leukemic agents given as post-transplant maintenance therapy (e.g., subcutaneous or oral 5-azacytidine or FLT3 inhibitors for maintenance)
* Active acute graft versus host disease (GVHD) grade II or higher
* Active chronic GVHD that is extensive
* Concurrent use of systemic immune suppressive other than calcineurin inhibitors and sirolimus
* Active uncontrolled systemic fungal, bacterial or viral infection
* Symptomatic or uncontrolled arrhythmias
* Significant active cardiac disease within the previous 6 months, including: New York Heart Association (NYHA) class III or IV congestive heart failure; unstable angina or angina requiring surgical or medical intervention, and/or; myocardial infarction
* Known active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Prior history of solid tumor unless the subject has been free of the disease for >= 1 year; however, subjects with the following history/concurrent conditions are allowed: basal or squamous cell carcinoma of the skin; carcinoma in situ of the cervix; carcinoma in situ of the breast; incidental histologic finding of prostate cancer (T1a or T1b using the tumor, node, metastasis [TNM] clinical staging system)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betul Oran, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were registered at MD Anderson Cancer Center.
Groups:
- Cohort 1: Relapsed Leukemia Post-transplant: Patients with morphological relapse for AML and MDS at least 90 days post-transplant.
  MDS patients: Re-appearance of dysplastic changes in the bone marrow, with or without increase in bone marrow blast count, which is pathologically consistent with myelodysplastic syndrome.
  AML patients:
  Bone marrow blast count >/= 5%.
- Cohort 2: MRD(Minimal Residual Disease) Post-transplant: Cohort 2: Persistence or reappearance of minimal residual disease by flow cytometry or cytogenetic or molecular testing while being in morphological remission after allogeneic stem cell transplantation.
- Cohort 3: Maintenance Treatment Post-transplant: Cohort 3: High risk AML and MDS patients who are in complete remission morphologically with no evidence of minimal residual disease by flow cytometry or cytogenetic or molecular testing after allogeneic stem cell transplantation.
Period: Overall Study
Arm/Group | Cohort 1: Relapsed Leukemia Post-transplant | Cohort 2: MRD(Minimal Residual Disease) Post-transplant | Cohort 3: Maintenance Treatment Post-transplant
Started | 13 | 18 | 24
Completed | 13 | 17 | 24
Not Completed | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Relapsed Leukemia Post-transplant | Cohort 2: MRD(Minimal Residual Disease) Post-transplant | Cohort 3: Maintenance Treatment Post-transplant | Total
Number analyzed (Participants) | 13 | 18 | 24 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 13 | 31
  >=65 years | 5 | 8 | 11 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 11 | 27
  Male | 8 | 7 | 13 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 2 | 7
  Not Hispanic or Latino | 9 | 17 | 22 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 18 | 24 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieved Complete Response (CR)
Description: Complete remission (CR): Bone marrow with </= 5% bone marrow blasts with normal maturation of all cell lines in the absence of extramedullary disease in addition to a peripheral blood granulocyte count >/= 1 X 10^9/L and a platelet count >/= 100 x 10^9 /L.
Time Frame: Within the first 6 cycles, up to 168 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Relapsed Leukemia Post-transplant | Cohort 2: MRD(Minimal Residual Disease) Post-transplant | Cohort 3: Maintenance Treatment Post-transplant
Number analyzed (Participants) | 13 | 18 | 24
Participants | 3 | 9 | 16

2. Secondary Outcome: Overall Survival (OS)
Description: Number of participants that are alive 1 year after study enrollment.
Time Frame: At 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Relapsed Leukemia Post-transplant | Cohort 2: MRD(Minimal Residual Disease) Post-transplant | Cohort 3: Maintenance Treatment Post-transplant
Number analyzed (Participants) | 13 | 18 | 24
Participants | 12 | 12 | 10

3. Secondary Outcome: Disease-free Survival
Description: Number of participants that are disease free and alive 1 year after study enrollment.
Time Frame: At 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Relapsed Leukemia Post-transplant | Cohort 2: MRD(Minimal Residual Disease) Post-transplant | Cohort 3: Maintenance Treatment Post-transplant
Number analyzed (Participants) | 13 | 18 | 24
Participants | 5 | 7 | 20

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cohort 1: Relapsed Leukemia Post-transplant | Cohort 2: MRD(Minimal Residual Disease) Post-transplant | Cohort 3: Maintenance Treatment Post-transplant
All-Cause Mortality (participants affected / at risk) | 1/13 | 6/18 | 14/24
Serious Adverse Events (participants affected / at risk) | 9/13 | 11/18 | 12/24
Other Adverse Events (participants affected / at risk) | 3/13 | 8/18 | 10/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Relapsed Leukemia Post-transplant (N=13) | Cohort 2: MRD(Minimal Residual Disease) Post-transplant (N=18) | Cohort 3: Maintenance Treatment Post-transplant (N=24)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 9 (10) | 11 (41) | 12 (50)
Platelet count decreased (Investigations) | 6 (6) | 6 (13) | 6 (6)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 6 (6) | 10 (13) | 9 (12)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Relapsed Leukemia Post-transplant (N=13) | Cohort 2: MRD(Minimal Residual Disease) Post-transplant (N=18) | Cohort 3: Maintenance Treatment Post-transplant (N=24)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 2 (7)
Anemia (Blood and lymphatic system disorders) | 3 (6) | 7 (14) | 5 (7)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (7) | 3 (3) | 2 (2)
Gallbladder infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 5 (7)
Nausea (Gastrointestinal disorders) | 2 (5) | 5 (5) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 5 (48) | 9 (56)
Platelet count decreased (Investigations) | 2 (8) | 8 (70) | 10 (76)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (3) | 4 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 1 (6) | 7 (65) | 9 (164)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 3 (3) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (9)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT02684162/Prot_SAP_001.pdf